CLINICAL TRIAL: NCT05834257
Title: Study on the Modulation of Inflammation by Crystalloid Fluids in Cardiac Surgery Patients
Brief Title: Crystalloid Fluids and Cardiac Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of participants
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15.167
Record Dates: First submitted 2023-04-04; First posted 2023-04-28 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Surgery-Complications
Keywords: cardiac surgery; renal failure
MeSH Terms: conditions — Renal Insufficiency | interventions — Saline Solution; Plasmalyte A

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Normal Saline (Experimental): 5 Cardiac surgery patients admitted to the intensive care units will receive, following consent and randomisation, Normal Saline as resuscitation fluid. 50mL of blood will be withdrawn before surgery and 24 hours after for each patient in order to isolate neutrophils and monocytes. Plasma will be preserved for future cytokines characterization.
  Interventions: Procedure: Normal Saline for fluid resuscitation
- PlasmaLyte (Experimental): 5 Cardiac surgery patients admitted to the intensive care units will receive, following consent and randomisation, PlasmaLyte as resuscitation fluid. 50mL of blood will be withdrawn before surgery and 24 hours after for each patient in order to isolate neutrophils and monocytes. Plasma will be preserved for future cytokines characterization.
  Interventions: Procedure: PlasmaLyte for fluid resuscitation
- Ringer's Lactate (Experimental): 5 Cardiac surgery patients admitted to the intensive care units will receive, following consent and randomisation, Ringer's lactate as resuscitation fluid. 50mL of blood will be withdrawn before surgery and 24 hours after for each patient in order to isolate neutrophils and monocytes. Plasma will be preserved for future cytokines characterization.
  Interventions: Procedure: Ringer's Lacatate for fluid resusciation

INTERVENTIONS:
Procedure: Normal Saline for fluid resuscitation — Fluid resuscitation is a critical and essential part in cardiac surgery procedures. Patients randomized for this arm will be submitted to Normal Saline infusion (as clinically prescribed).
  Arms: Normal Saline
Procedure: PlasmaLyte for fluid resuscitation — Fluid resuscitation is a critical and essential part in cardiac surgery procedures. Patients randomized for this arm will be submitted to PlasmaLyte infusion (as clinically prescribed).
  Arms: PlasmaLyte
Procedure: Ringer's Lacatate for fluid resusciation — Fluid resuscitation is a critical and essential part in cardiac surgery procedures. Patients randomized for this arm will be submitted to Ringer's Lactate infusion (as clinically prescribed).
  Arms: Ringer's Lactate

SUMMARY:
All cardiac patients admitted to the intensive care unit after surgery received crystalloid fluids as standard care procedure. 3 crystalloid fluids can be used during their stay: Normal Saline, PlasmaLyte or Ringer's Lactate. They differ in their respective composition, mainly in chloride and sodium concentrations. Inflammatory consequences of the crystalloid fluids used in this population are unknown. The investigators plan to evaluate which one of the three fluids mentioned above is advantageous in cardiac surgery patients with regards to reduced rate of infection and renal failure.

DETAILED DESCRIPTION:
Inflamed patients admitted to the intensive care unit after cardiac surgery received large volumes of crystalloid fluids as standard care procedure. The goal is to control the balance between the initial pro-inflammatory phase and the subsequent/compensatory anti-inflammatory phase, the later being associated to immune fatigue and the apparition or re-activation of infections. Infectious complications are responsible for the increased rate of morbidity and mortality in this cardiac surgery population. The inflammatory impacts of each of the crystalloid fluids administered to the patient are still ill-defined and represent an opportunity to better control the hyperinflammation and/or immunosuppression often observed following cardiac surgery. Hence, the investigators will evaluate the activation of the immune system following crystalloid fluid (either Normal saline (NS), PlasmaLyte (PL) or Ringer's Lactate (RL)) administration in this population with regard to one recurrent clinical issue, i.e renal failure.

The hypothesis is that LR is less ''immuno-activator'' on monocytes than NS and PL. The objectives are: 1-evaluate the inflammatory profiles of each of the crystalloid fluids in consent cardiac surgery patients during their stay in the intensive care unit by studying white blood cell phenotypes and inflammatory cytokines present in plasma and 2-evaluate the impacts of crystalloid fluids in vitro using white blood cell from cardiac surgery patients obtained before surgery.

ELIGIBILITY:
Inclusion Criteria:

* patient for coronary artery bypass surgery with CPB (Cardiopulmonary bypass)

Exclusion Criteria:

* use of immunomodulating medication 6 months before surgery
* chemiotherapy/radiotherapy 6 months before surgery
* history of neoplasia
* auto-immune disorders
* pregnancy
* severe infection 1 month before surgery
* renal/hepatic failure
* left ventricular ejection fraction <40%
* hepatitis C or HIV
* symptomatic peripheral vascular diseases
* chronic obstructive pulmonary disease
* cerebrovascular accident
* hemoglobin <90g/L
* leukocytes <6 or >12x10e6/L

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-03-31 (Actual); Primary Completion 2025-02-19 (Actual); Study Completion 2025-02-19 (Actual)

PRIMARY OUTCOMES:
Change in monocyte phenotype before and after cardiac surgery | 24 hours
  Using white blood cells from patients, the investigators will evaluate CD14/16 expression on monocytes by flow cytometry before and after infusion of crystalloid fluids. Results will be presented as percentage of positive cells.

SECONDARY OUTCOMES:
Sequential Organ Failure Assessment (SOFA) score after cardiac surgery | 48 hours
  will be evaluated by the clinical team. Scale range is 0 (normal, best outcome) to 24 (abnormal, worse outcome).
Length of stay in intensive care unit after cardiac surgery | up to 4 weeks
  will be monitored by the clinical team

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François Cailhier, MD, Principal Investigator — CRCHUM
Locations (1):
- Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
as mentioned below. Patient names won't be available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Following completion of the study and upon demand
Access Criteria: reasonable request